CLINICAL TRIAL: NCT00611598
Title: DNA Repair and Genetic Susceptibility to Lung Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 03-003
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Lung Cancer; Single Primary Lung Cancer; Second Primary Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * 30 ml. Blood in heparinized, green top tubes.
  * Fresh tumor or normal tissue, when available.
  * Tissue or cells from routine bronchoscopy, when available.

GROUPS / COHORTS (2):
- 1: second primary lung cancer
  Interventions: Other: Blood draw and Questionnaires
- 2: single primary lung cancer
  Interventions: Other: Blood draw and Questionnaires

INTERVENTIONS:
Other: Blood draw and Questionnaires — Pt will have three green top tubes of blood drawn. The questionnaire will be filled out by the study subject. This may be completed at home and mailed in a provided stamped addressed envelope if the patient prefer, or obtained by phone interview with a research assistant.
  Groups: 1
Other: Blood draw and Questionnaires — Pt will have three green top tubes of blood drawn. The questionnaire will be filled out by the study subject. This may be completed at home and mailed in a provided stamped addressed envelope if the patient prefer, or obtained by phone interview with a research assistant.
  Groups: 2

SUMMARY:
The purpose of this study is to help us better understand the cellular changes that may lead to the development of lung cancer. We want to compare people with a second primary lung cancer with those who have only a first primary lung cancer. We hope to use the information obtained in this study as the basis for future studies and will not regard the results from this study as final.

We will analyze your blood cells and DNA to measure the changes in several genes that we believe may be involved in lung cancer. We also want to evaluate the capacity for your DNA to repair itself.

ELIGIBILITY:
Inclusion Criteria:

* Cases will be eligible for inclusion if:
* They have been diagnosed with a second primary lung cancer, and
* They speak English or a language for which we have a translated consent form, and
* They understand and agree to sign informed consent, and
* They agree to give us a blood sample, and
* They agree to give us a tissue sample when part of normal clinical procedures, and
* They agree to complete the study questionnaires, and
* They agree to have their pathology information reviewed. This could include biopsy specimens.

Controls will be eligible for inclusion if

* They have been diagnosed with a first primary lung cancer, and
* They speak English or a language for which we have a translated consent form, and
* They understand and agree to sign informed consent, and
* They agree to give us a blood sample, and
* They agree to give us a tissue sample when part of normal clinical procedures, and
* They agree to complete the study questionnaires,
* They agree to have their pathology information reviewed. This will could include biopsy specimens.

Exclusion Criteria:

* Subjects who do not meet the inclusion criteria as either cases or controls will not be eligible for this study.
* Control subjects who have a history of another cancer, other than nonmelanoma skin cancer or a first primary lung cancer, will not be eligible for this study.
* Control subjects who otherwise meet the eligibility requirements above but who have had chemotherapy and/or are currently being treated with chemotherapy will be excluded from the functional assay, but not from the genotyping.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: MSKCC Clinic
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2003-02-11 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
To conduct a pilot study of the role of DNA repair in lung cancer subjects with high genetic risk - those with a second primary lung cancer - compared to subjects with only one lung cancer. | conclusion of the study

SECONDARY OUTCOMES:
To determine the association between cellular DNA repair and genetic alterations in DNA repair and associated pathways. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Irene Orlow, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org